CLINICAL TRIAL: NCT03430414
Title: Transcriptome Analysis of Stored Biopsy Samples in Clinically Precisely Phenotyped Therapy-responders Versus Non-responders Diagnosed With Antibody Mediated Rejection
Brief Title: Analysis of Biopsies With Antibody Mediated Rejection According to the Therapy Response
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Thomas Mueller (Other)
Responsible Party: Sponsor-Investigator, Thomas Mueller, Professor, University of Zurich
Organization: University of Zurich (Other)
Other Study IDs: BASEC-Nr. 2017-02130
Record Dates: First submitted 2018-02-05; First posted 2018-02-12 (Actual); Last update posted 2018-02-12 (Actual); Status verified 2018-02

CONDITIONS: Antibody-mediated Rejection
MeSH Terms: interventions — Transcriptome

STUDY DESIGN:
Observational Model: Other | Time Perspective: Retrospective
Biospecimen Retention: RNA Analysis of Formalin Fixed Paraffin Embedded biopsies
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Therapy Responders
  Interventions: Diagnostic Test: Transcriptome Analysis
- Non-Responders
  Interventions: Diagnostic Test: Transcriptome Analysis

INTERVENTIONS:
Diagnostic Test: Transcriptome Analysis — Transcriptome Analysis of Formalin Fixed Paraffin Embedded biopsies

SUMMARY:
In adult kidney transplant recipients a therapy-responder and non-responder phenotype by antibody mediated rejection will be precisely defined according to clinical and histological characteristics such as creatinine, proteinuria and Banff-classification. Twenty-five patients will be selected each in the therapy-responder and non-responder group. Their stored Formalin Fixed Paraffin Embedded (FFPE) biopsies will be (re)-classified according to the most recent Banff classification. Using Nanostring Technology the gene transcription of therapy-responders versus non-responders will be analyzed and compared to serological and clinical parameters.

ELIGIBILITY:
Inclusion Criteria:

* Kidney transplant patients at the University Hospital of Zurich between 01.01.2008 - 31.12.2016 with histologically suspected or confirmed ABMR
* Written consent for further use of data for research purposes

Exclusion Criteria:

* Age at transplantation < 18 years
* Combined organ transplantation (incl. Kidney-Pancreas, Kidney-Liver, Kidney-Heart)
* Incomplete laboratory and/or clinical data
* Recurrence of the initial disease
* Insufficient Biopsy Material for NanoString Analysis
* Documented refusal of further data analysis for research purpose

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All ABMR cases in patients who received a kidney transplant between 01.01.2008 - 31.12.2016 will be pre-screened. As an approximate number of 90 kidney transplantations are performed per year at the University Hospital of Zürich, a total of approximately 810 patients will be available for analysis. Yet, according to the inclusion/exclusion criteria we estimate roughly 50 patients to be finally recruited for analysis. Since we estimate a consent rate of about 50%, we will roughly contact 100 patients. A subset of 25 responders and 25 non-responders according to the clinical course will be identified for further analysis
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2018-02-15 (Estimated); Primary Completion 2018-03-01 (Estimated); Study Completion 2018-04-30 (Estimated)

PRIMARY OUTCOMES:
Transcriptome | 02.15.2018-03.01.2018
  mRNA

REFERENCES:
- [Derived] Sazpinar O, Gaspert A, Sidler D, Rechsteiner M, Mueller TF. Histologic and Molecular Patterns in Responders and Non-responders With Chronic-Active Antibody-Mediated Rejection in Kidney Transplants. Front Med (Lausanne). 2022 Apr 29;9:820085. doi: 10.3389/fmed.2022.820085. eCollection 2022. PMID 35573002